CLINICAL TRIAL: NCT04473209
Title: The Effect of Non-surgical Periodontal Therapy on Serum Resistin Level in Chronic Periodontitis Patients With or Without Type 2 Diabetes Mellitus
Brief Title: Serum Resistin Level Following Non-surgical Periodontal Therapy in Diabetic Patients With Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Weam Ahmed Elbattawy, Dr. Principal Investigator, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: version 1
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Intervention Model Description: group1: diabetic patients with chronic periodontitis group2: non diabetic patients with chronic periodontitis
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- diabetic group (Active Comparator): diabetic patients with chronic periodontitis
  Interventions: Procedure: non-surgical periodontal therapy
- non-diabetic group (Active Comparator): non diabetic patients with chronic periodontitis
  Interventions: Procedure: non-surgical periodontal therapy

INTERVENTIONS:
Procedure: non-surgical periodontal therapy — supra and subgingival debridement

SUMMARY:
non-surgical periodontal debridement was performed for diabetic patients with chronic periodontitis as well as for non-diabetic patients but also with chronic periodontitis. Serum resistin level was assessed in the two groups before and after periodontal therapy and also was compared to a healthy control group.

DETAILED DESCRIPTION:
Background: Resisitin is a recognized marker for chronic inflammatory conditions that could be directly linked with type 2 diabetes mellitus. The aim of this study was to assess serum resistin level in type 2 diabetic patients with chronic periodontitis.

Methods: Forty individuals were recruited in this study and were divided into three groups, diabetic group consisted of 15 diabetic patients (type 2 diabetes mellitus) with moderate to severe chronic periodontitis, non-diabetic group consisted of 15 non-diabetic patients with moderate to severe chronic periodontitis and healthy group consisted of 10 non-diabetic individuals with healthy periodontium. Non-surgical periodontal therapy with supra and subgingival debridement was performed for the diabetic and non-diabetic groups. Pocket depth, clinical attachment level, plaque index, gingival index, serum Resistin and high sensitivity C-Reactive Protein assay were recorded for both groups before and after treatment, while HbA1c was recorded for the diabetic group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with moderate to severe chronic periodontitis.
* Presence of a minimum of 15 natural teeth
* Presence of at least four teeth with one or more sites with probing pocket depth (PPD) ≥5mm and clinical attachment level (CAL) ≥4mm
* agreement to participate in the study and sign a written informed consent

Exclusion Criteria:

* Patients who received any periodontal treatment or professional scaling and root planing of the teeth for at least 6 months prior to the study initiation
* A history of antibiotics therapy and anti-inflammatory drugs within the previous 6 months
* Pregnancy or use of contraceptives or any medication related to diabetes
* former or current smokers ˂ 5 years.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
serum resistin | 3 months
  ng/ml

SECONDARY OUTCOMES:
C-reactive protein | 3 months
  μg/mL
probing pocket depth | 3 months
  mm
clinical attachment loss | 3 months
  mm

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt